CLINICAL TRIAL: NCT00940043
Title: Monitoring of Women With Preterm Premature Rupture of Membranes (PPROM) Between 28 and 33 Weeks of Gestation With Repetitive Immunochromatographic Bedside Test to Detect Inflammatory Protein in Vaginal Secretions.
Brief Title: Monitoring of the Inflammatory Response of Patients With Premature Rupture of Membranes With Bedside Tests
Acronym: EFFARM
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, DR, Université de Sherbrooke
Other Study IDs: 08-072
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Premature Rupture of Fetal Membranes
Keywords: bedside test; interleukins; inflammation; vaginal secretions
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — vaginal secretions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rupture of fetal membranes: women with rupture of fetal membranes before onset of labor

SUMMARY:
Prematurity represents 8% of birth and it is one of the leading causes of infant complications. The preterm premature rupture of membranes (PPROM) represents one-third of preterm birth and the rupture of membranes increase the risk of fetal exposition to infection which could lead to neurological sequels. Classic management of women with PPROM before 32SA is based on the extension of the pregnancy with the risk of adding complications like a secondary infection. Moreover, different studies have shown that fetal infection could be one of the most important risk factor for subsequent neurological complications. However, it is difficult to know if it is better to extend the pregnancy to gain in maturity or to arrest the pregnancy to avoid the risk of intrauterine infection. The research objective is to suggest a new strategy to manage women with PPROM. With this new strategy, the investigators seek to extend pregnancy as much as possible but the investigators would like to give birth before the intrauterine infection. The investigators suggest detecting protein associate with neurological complications of preterm child in the amniotic liquid found in the vagina of the mother. A positive test will lead to the delivery of the newborn before its infection. The hypothesis is that it is possible to study changes in the inflammatory status of patients who presented an PPROM from repeated detection of interleukins in vaginal secretions.

DETAILED DESCRIPTION:
Preterm premature rupture of the membranes (PPROM) represents one-third of preterm births and is the leading cause of perinatal mortality and morbidity. During the latency period, several events such as the ascent of pathogenic microorganisms from the lower genital area could create complications which may culminate in cerebral palsy. Avoiding intrauterine infection appears as one of the most important objective in the PPROM management. Most authors propose the conservative management of women with PPROM, associating antibiotic therapy to corticosteroid administration in patients with PPROM before 30 to 32 weeks. The main benefit of conservative management is prolonging pregnancy, but the benefit must be balanced with the risks of fetal complications. In an effort to diminish the risks of infection linked to a longer latency period, several authors have proposed intentional delivery after PPROM.

The primary objective is the comparison between the results of IMMUNOCHROMATOGRAPHY tests done at the bedside of the patient and the ELISA tests performed in the laboratory.

The secondary outcome is the description of the inflammatory status following a rupture of membranes at term and during labor.

Vaginal secretions samplings are perform after premature rupture of membranes and during labor. The bedside test is performing immediately after sampling and the rest of the sampling is frozen. ELISA assays will be performed on these samples.

ELIGIBILITY:
Inclusion Criteria:

* Women with a single fetus and hospitalized for a rupture of membranes at term or before term.

The criteria for diagnosis of rupture of membranes is based on clinical and biochemical tests, including Fern test and Actim PROM test

Exclusion Criteria:

* Twin pregnancies, patients in labor, the presence of medical complications which exclude expectant management including abruptio placentae, preeclampsia or eclampsia and fetal death.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women hospitalized for premature rupture of membranes at the CHUS
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
comparison between the results of the bedside test and the ELISA tests performed in the laboratory | after rupture of membranes

SECONDARY OUTCOMES:
description of the inflammatory status following a rupture of membranes at term and during labor | after rupture of membranes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Sherbrooke
Locations (1):
- Centre hospitalier de l'Université de Sherbrooke, Sherbrooke, Quebec, Canada